CLINICAL TRIAL: NCT05128110
Title: Study of Hemostasis During the Atrial Fibrillation Ablation Procedure
Acronym: EHPAFAVE
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7717
Record Dates: First submitted 2021-10-06; First posted 2021-11-19 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-10

CONDITIONS: Hemostasis
Keywords: Atrial fibrillation; Ablation; ACT; Heparin; Direct oral anticoagulant
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anticoagulation monitoring is done by monitoring the ACT (Activated Clotting Time) with an objective greater than 300 s. Until now, treatment with direct oral anticoagulant (for the prevention of thromboembolic events of atrial fibrillation) was interrupted a few days before the procedure in order to limit the risk of per-procedural bleeding. However, 3 recent randomized studies concerning the 3 DOACs available suggest that treatment should not be interrupted during the entire operative period. The operation therefore takes place under double anticoagulation with a direct oral anticoagulant and unfractionated heparin. Under these conditions, ACT monitoring can no longer be considered a reliable means of measuring the level of anticoagulation. It was therefore necessary to explore the hemostasis of these patients in a broad way in order to avoid any risk of overdose of UFH (Unfractionated Heparin) during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years-old
* with an atrial fibrillation
* Operated for an atrial fibrillation procedure in the University hospital of Strasbourg
* Without interruption of the direct oral anticoagulant
* For whom extended biological assessment has been made in routine practice

Exclusion Criteria:

* Patients who refused the use of their data for this study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient with an atrial fibrillation, perated for an atrial fibrillation procedure in the University hospital of Strasbourg and without interruption of the direct oral anticoagulant
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Study of hemorrhagic and thrombotic complications and correlation with the various laboratory tests | Files analysed retrospectively from January 01, 2019 to December 31, 2019 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Charles-Ambroise TACQUARD, MD, Principal Investigator — Service d'Anesthésie et Réanimation chirurgicale - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service d'Anesthésie et Réanimation chirurgicale - Hôpitaux Universitaires de Strasbourg, Strasbourg, France